CLINICAL TRIAL: NCT02168673
Title: Modulation of Genes Responsible for Cilia Length by Exposure to Cigarette Smoke
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1102011549
Record Dates: First submitted 2014-06-10; First posted 2014-06-20 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: COPD; Smoking
Keywords: COPD; Cigarette Smoke; Smoker; Nonsmoker; ODF2; Cilia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Cigarette Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and cells obtained from the study may be kept for future genetic studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Healthy non-smokers
- Group 2: Healthy non-smokers

SUMMARY:
Cigarette smoking is the major risk factor for developing chronic obstructive pulmonary disease (COPD). Patients with COPD have difficulty clearing mucus and debris from their airways. Even smokers who have not developed COPD may have difficulty clearing the airways. This is partly because smoking impairs the function of cilia, tiny hairs lining the airways that sweep out mucus to keep the airways clean. The investigators have found that smoking reduces the length of cilia, which may contribute to the worsened cilia function in smoking and COPD. This is true even in smokers who show no signs of lung disease. The investigators believe that smoking affects levels of genes in lung cells, resulting in shorter cilia.

DETAILED DESCRIPTION:
In this study, we will use bronchoscopy (inserting a scope into the lungs) to obtain lung cells by brushing cells from the airways and we will study genes that may be related to cilia length. Our goals are (1) to prove that exposure to cigarette smoke results in shorter cilia, (2) to learn which specific genes control cilia length, and (3) to learn how smoking affects the gene ODF2 and what effect this has on cilia. Understanding how smoking affects cilia may help us identify new ways to treat patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Must be capable of providing informed consent
* Males and females, age 18 or older
* Nonsmoking, validated by venous carboxyhemoglobin and urine nicotine and cotinine within range for nonsmoker without smoke exposure, matched with smoker group by age, sex, ethnic/racial group
* Good overall health without history of chronic lung disease, including asthma, and without recurrent or recent (within 3 months) acute pulmonary disease
* Normal physical examination
* Normal routine laboratory evaluation, including general hematologic studies, general serologic/immunologic studies, general biochemical analyses, and urine analysis
* Negative HIV, hepatitis B and C serology
* Normal chest X-ray (PA and lateral)
* Normal electrocardiogram
* Females - not pregnant
* No history of allergies to medications to be used in the bronchoscopy procedure
* Not taking any medications relevant to lung disease or having an effect on the airway epithelium
* Willingness to participate in the study

Exclusion Criteria:

* Unable to meet the inclusion criteria
* Pregnancy
* Current active infection or acute illness of any kind
* Habitual use of drugs and/or alcohol within the past six months (Acceptable: -Marijuana one time in three months; average of two alcoholic beverages per day; drug and/or alcohol abuse is defined as per the DSM-IV Substance Abuse Criteria)
* Evidence of malignancy within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will involve healthy nonsmokers and healthy smokers.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Evidence that exposure to cigarette smoke will result in shorter cilia length in human airway epithelial | One Year
  Cilia length will be measured using three preparation techniques: air-dried cytospins, detached cilia on cytospins, and mounted hydrated aliquots of cells.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College and Weill Cornell Medical Center, Department of Genetic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided